CLINICAL TRIAL: NCT00000959
Title: Prophylaxis Against Tuberculosis (TB) in Patients With Human Immunodeficiency Virus (HIV) Infection and Suspected Latent Tuberculous Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: CPCRA 005; 11557 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Tuberculosis
Keywords: Tuberculosis; Isoniazid; Pyridoxine; AIDS-Related Opportunistic Infections; Drug Evaluation; Acquired Immunodeficiency Syndrome; Antitubercular Agents
MeSH Terms: conditions — HIV Infections; Tuberculosis; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome | interventions — Isoniazid; Pyridoxine

INTERVENTIONS:
Drug: Isoniazid
Drug: Pyridoxine hydrochloride

SUMMARY:
To evaluate the safety and effectiveness of a 6-month course of isoniazid ( INH ) in the prevention of clinical tuberculosis in anergic (having diminished or absent reactions to specific antigens) HIV-infected persons who are at high risk for tuberculous infection.

A substantial number of HIV-infected persons are anergic, and thus do not respond to the only currently available diagnostic tool for tuberculosis infection (that is, the PPD (purified protein derivative) skin test). Many of these anergic persons are, however, infected with Mycobacterium tuberculosis and eventually develop reactivation tuberculosis, causing both individual illness and spread of infection to others in the community. This study examines the possibility of using INH prophylaxis (that is, for prevention) in anergic HIV-infected patients at high risk for tuberculosis as a means of decreasing the sharp rise in the incidence of tuberculosis due to HIV infection. INH is inexpensive and relatively safe, and thus may demonstrate an acceptable risk/benefit ratio as a medication that can be given over a limited period of time to a population suspected of having, but not proved to have, M. tuberculosis infection. If this study shows INH to be safe and effective in this setting, it could have a major effect on public health in this country.

DETAILED DESCRIPTION:
A substantial number of HIV-infected persons are anergic, and thus do not respond to the only currently available diagnostic tool for tuberculosis infection (that is, the PPD (purified protein derivative) skin test). Many of these anergic persons are, however, infected with Mycobacterium tuberculosis and eventually develop reactivation tuberculosis, causing both individual illness and spread of infection to others in the community. This study examines the possibility of using INH prophylaxis (that is, for prevention) in anergic HIV-infected patients at high risk for tuberculosis as a means of decreasing the sharp rise in the incidence of tuberculosis due to HIV infection. INH is inexpensive and relatively safe, and thus may demonstrate an acceptable risk/benefit ratio as a medication that can be given over a limited period of time to a population suspected of having, but not proved to have, M. tuberculosis infection. If this study shows INH to be safe and effective in this setting, it could have a major effect on public health in this country.

Patients are placed by a random selection process in either the INH or placebo group. One group receives INH plus pyridoxine hydrochloride ( vitamin B6 ) daily for six months. Patients in the other group receive placebo plus vitamin B6 daily for six months.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Antiretroviral therapy.
* Pneumocystis carinii pneumonia prophylaxis.
* Treatment for acute opportunistic infections/malignancies.

Patients must have:

* Reasonably good health.
* Life expectancy of at least six months.
* Willing and able, in the clinician's opinion, to comply with the treatment and clinical management issues as outlined in the protocol.
* HIV infection.
* Signed informed consent.

Allowed:

* Participation in other clinical trials as long as there is no potential activity of other study drugs against M. tuberculosis, additive toxicities between study agents, or known possible drug interactions between study drugs.
* Must be in a high-risk group for Mycobacterium tuberculosis infection, including:
* foreign-born from countries with a high prevalence of M. tuberculosis infection; from medically underserved low-income populations (high-risk racial or ethnic minority populations such as African Americans, Hispanic / Latinos, Native Americans, and/or the homeless, unemployed, inner city residents); alcohol or injectable drug users; or residents or former residents of high-risk, long-term care or residential facilities (correctional or mental institutions, nursing homes).

Prior Medication:

Allowed:

* Previous treatment with quinolones/fluoroquinolones, aminoglycosides, or other agents with known or potential activity against M. tuberculosis.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Current active clinical tuberculosis, confirmed or suspected, or household contact with someone with active clinical tuberculosis.
* History of sensitivity/intolerance to the study medication.
* Evidence of peripheral neuropathy, i.e., signs or symptoms of paresis, paresthesias, neuromotor abnormalities, or neurosensory deficits of grade 3 or worse.
* Evidence of acute hepatitis.

Concurrent Medication:

Excluded:

-

Quinolones, fluoroquinolones, or aminoglycosides with antituberculous activity (may be used for up to 14 days for treatment of intercurrent infection). Other agents with known or potential antituberculosis activity should be avoided, including the following:

* Aminosalicylic acid salts, capreomycin, clofazimine, cycloserine, ethambutol, ethionamide, isoniazid, kanamycin, pyrazinamide, rifabutin, rifampin, streptomycin, or thiacetazone.

Prior Medication:

Excluded:

* Treatment for more than 1 month (continuous or cumulative) with drugs that have known or potential antituberculous activity, other than quinolones, fluoroquinolones, and some aminoglycosides.

Patients may not have:

* Current active clinical tuberculosis, confirmed or suspected, or household contact with someone with known active clinical tuberculosis.
* Evidence of peripheral neuropathy, i.e., signs or symptoms of paresis, paresthesias, neuromotor abnormalities, or neurosensory deficits of grade 3 or worse.
* Unable or unwilling to have current therapy and/or concomitant medications changed to avoid serious interaction with study medication.
* Documented history of a positive PPD skin test.
* Participation in other clinical trials in which there is potential activity of other study drugs against M. tuberculosis, additive toxicities between study agents, or known possible drug interactions between study drugs.

Alcohol or injectable drug users.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600
Dates: Study Completion 1996-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gordin F, Study Chair
Locations (14):
- United States (14):
  - UCLA Med Ctr, Los Angeles, California
  - Community Consortium of San Francisco, San Francisco, California
  - Denver CPCRA / Denver Public Hlth, Denver, Colorado
  - Hill Health Corp, New Haven, Connecticut
  - Wilmington Hosp / Med Ctr of Delaware, Wilmington, Delaware
  - Veterans Administration Med Ctr / Regional AIDS Program, Washington D.C., District of Columbia
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Louisiana Comm AIDS Rsch Prog / Tulane Univ Med, New Orleans, Louisiana
  - Comprehensive AIDS Alliance of Detroit, Detroit, Michigan
  - North Jersey Community Research Initiative, Newark, New Jersey
  - Addiction Research and Treatment Corp, Brooklyn, New York
  - Clinical Directors Network of Region II, New York, New York
  - Harlem AIDS Treatment Group / Harlem Hosp Ctr, New York, New York
  - Bronx Lebanon Hosp Ctr, The Bronx, New York

REFERENCES:
- [Background] Gordin FM, Matts JP, Miller C, Brown LS, Hafner R, John SL, Klein M, Vaughn A, Besch CL, Perez G, Szabo S, El-Sadr W. A controlled trial of isoniazid in persons with anergy and human immunodeficiency virus infection who are at high risk for tuberculosis. Terry Beirn Community Programs for Clinical Research on AIDS. N Engl J Med. 1997 Jul 31;337(5):315-20. doi: 10.1056/NEJM199707313370505. PMID 9233868